CLINICAL TRIAL: NCT03748667
Title: Diagnostic Accuracy of Deep Submucosal Invasion: White Light Endoscopy vs Invasive Pattern Based on NBI/BLI ± Chromoendoscopy
Brief Title: Accuracy for Predicting Deep Submucosal Invasion
Acronym: NBIBLI
Status: Completed | Type: Observational
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Collaborators: Hospital Universitario La Fe (Other); Hospital Clínico Universitario Lozano Blesa (Other); University of North Carolina, Chapel Hill (Other); Hospital Clinic of Barcelona (Other); National Cancer Center, Japan (Other Government); Germans Trias i Pujol Hospital (Other); Hospital Universitario 12 de Octubre (Other); Hospital Universitario Ramon y Cajal (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Comarcal de Alcañiz (Unknown); Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Ignasi Puig, Gastroenterology consultant, MD, PhD, Althaia Xarxa Assistencial Universitària de Manresa
Other Study IDs: CEIC 18/53
Record Dates: First submitted 2018-11-13; First posted 2018-11-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Colorectal Polyp
Keywords: Endoscopy; Colonoscopy; Invasive pattern; Polypectomy; NBI; BLI; Deep submucosal invasion; JNET; Kudo pit pattern
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Paraffin blocks of colorectal polyps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with colorectal polyps: Patients with non-pedunculated type 0 lesions in Paris classification (not obvious cancers) larger than 10 mm
  Interventions: Diagnostic Test: White light endoscopy (WLE); Diagnostic Test: NBI/BLI +/- chromoendoscopy (NBIBLI +/- CE)

INTERVENTIONS:
Diagnostic Test: White light endoscopy (WLE) — Subjective endoscopic assessment of deep submucosal invasion based on the presence of gross morphological malignant features, morphology and size.
Diagnostic Test: NBI/BLI +/- chromoendoscopy (NBIBLI +/- CE) — Endoscopic assessment of deep submucosal invasion with NBI and dual focus/magnification or BLI and magnification. In the case of demarcated areas or JNET 2B, Kudo pit pattern assessment with crystal violet will be performed.

SUMMARY:
The main aim of this study is to determine whether the assessment of the invasive pattern based on NBI with dual focus/magnification or BLI with magnification ± chromoendoscopy (NBI+CE) for predicting deep invasion is significantly more accurate than the assessment based on white light endoscopy (WLE), carried out by trained endoscopists.

DETAILED DESCRIPTION:
A video with the lesion assessment, without any data on the patient, will be recorded in a device connected to the processor provided by the Principal Investigator. The name of the file will be the record ID. All the lesions will be tested by the same endoscopist in vivo and an assistant will fulfill the data collection sheet during the colonoscopy.

First, the lesions will be cleaned and observed in a stable position. Size, location, morphology, demarcated areas, and gross morphological malignant features will be evaluated. Based on these WLE characteristics, a deep invasion prediction will be performed (control test). Second, the lesion will be assessed using NBI with near focus or magnification or BLI with magnification. A second cleaning with pronase (or N-acetylcysteine if pronase is not available) if the surface cannot be clearly observed because of the presence of mucus or if crystal violet is going to be used. Crystal violet 0.05% will be used in case of polyps type 2B in the JNET classification or lesions with a demarcated area. A non-traumatic catheter (or spray catheter) will be used to spray the crystal violet over the lesion. A final prediction of deep invasion will be performed for NBI or BLI ± CE (test evaluated).

The use of a cap to observe the bottom of the lesion, fix the lesion close to the endoscope or to observe the lesion underwater immersion is strongly recommended.

The resection technique will be decided upon according to the local experience. In case of endoscopy resection (cold snare, EMR, ESD, full thickness), lesions will be removed via the anus (not through the endoscopy channel) in order to preserve their integrity. Although EMR is performed, if possible, lesions will be referred to the pathologist well oriented and pinned out on a cork based, as is standard procedure in ESD.

In order to ensure that endoscopic assessment is performed before the histology evaluation, both diagnostic assessments (control test and test evaluated) will be recorded on the REDCap database on the day of the colonoscopy. REDCap records the time and date of all changes in the variables' results. The remaining variables (demographic data, etc.) will be recorded on the data collection sheet and copied later into REDCap.

Videos of the lesion assessments will be sent to the Principal Investigator. Centralized visualization will be conducted to detect protocol violations and to exclude lesions from the study.

A blinded histology assessment will be conducted by the local pathologist and if a carcinoma with submucosal invasion is diagnosed, histology slides will be referred for an additional blinded and centralized histology evaluation at the end of the study.

Pathologists participating in the histological phase will assess all the slides with submucosal invasion and will collect the histological factors associated with lymph node metastasis.

Finally, investigators participating in the translational phase will refer paraffin blocks of 10 lesions of each JNET category (2A, 2B and 3) for genetic tests (sequencing of a panel of 45 genes and analysis of alterations in the number of copies of the genome).

ELIGIBILITY:
Inclusion criteria:

* Non-pedunculated type 0 lesions in Paris classification (not obvious cancers)
* Lesions larger than 10 mm

Exclusion criteria are:

* Lesions assessed as JNET 1 by the endoscopist or serrated by the pathologist
* Previous biopsy or resection attempt
* Previous CT, MR or USE
* Unavailable histology
* Inflammatory bowel disease
* Informed consent not obtained
* Protocol violation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients > 18 years old who undergo a colonoscopy for any reason
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
The presence or absence of deep invasion according to the control test (WLE) | One day
  Deep invasion will subjectively be diagnosed based on the presence of gross morphological malignant features, morphology and size. No single malignant feature, specific morphology or size is required. The importance given to each criterion and the final diagnosis of deep invasion is based on the personal experience of the endoscopist.
The presence or absence of deep invasion according to the test evaluated (NBI/BLI +/- CE) | One day
  Deep invasion will be diagnosed in case of:
  * JNET type 3 or
  * JNET 2B + Kudo Vn pit pattern or
  * JNET 2B and Kudo Vi pit pattern fulfilling all the following criteria: severe Kudo Vi pit pattern + presence of a demarcated area + size (demarcated area) >6 mm for PG or 3 mm for NPG.
The presence or absence of deep invasion according to the gold standard (histology) | One day
  Deep invasion will be diagnosed if sm invasion ≥1000 μm is measured according to the Japanese guidelines by the central pathologists.

SECONDARY OUTCOMES:
Presence of any genetic mutations | one day
  Sequencing of a panel of colorectal cancer genes: the 45 genes will be sequenced frequently mutated in colorectal cancer, through the protocols established in the center Executor: APC, TP53, FBXW7, SOX9, ATM, SMAD4, KRAS, PIK3CA, AMER1, FAT4, ARID1A, BRAF, NRAS, CTNNB1, TCF7L2, ERBB2, MET, EGFR, HRAS, SETD2, DLC1, CDKN2A, PTEN, ARID2, FAT1, POLE, POLD1, NOTCH1, BRCA2, LRP1B, KMT2C, KMT2D, DAPK1, CSMD1, MUC16, ADAMTS15, SYNE1, PCLO, ZFHX4, RYR3, RYR2, RELN, IRS2, GNAS, DMBT1.
Number of genome copies using SNP-arrays | one day
  Number of copies using SNP-arrays.

CONTACTS AND LOCATIONS:
Overall Officials: Ignasi Puig, MD, PhD, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa
Locations (14):
- United States (2):
  - San Francisco Veterans Affairs Medical Center. University of California, San Francisco, California
  - University of North Carolina, Chapel Hill, North Carolina
- National Cancer Center, Tokyo, Japan
- Spain (11):
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitari Germans Trias i Pujol (Can Ruti), Badalona, Catalonia
  - Hospital Clínic de Barcelona, Barcelona, Catalonia
  - Institut d'Investigacions Biomèdiques August Pi i Sunyer (IDIBAPS), Barcelona, Catalonia
  - Althaia. Xarxa Assistencial Universitària de Manresa, Manresa, Catalonia
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Comarcal de Alcañiz, Alcañiz, Teruel
  - Hospital Universitario y Politécnico de La Fe, Valencia, Valencia
  - Centro Médico Teknon, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Backes Y, Moss A, Reitsma JB, Siersema PD, Moons LM. Narrow Band Imaging, Magnifying Chromoendoscopy, and Gross Morphological Features for the Optical Diagnosis of T1 Colorectal Cancer and Deep Submucosal Invasion: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2017 Jan;112(1):54-64. doi: 10.1038/ajg.2016.403. Epub 2016 Sep 20. PMID 27644737
- [Background] Hayashi N, Tanaka S, Hewett DG, Kaltenbach TR, Sano Y, Ponchon T, Saunders BP, Rex DK, Soetikno RM. Endoscopic prediction of deep submucosal invasive carcinoma: validation of the narrow-band imaging international colorectal endoscopic (NICE) classification. Gastrointest Endosc. 2013 Oct;78(4):625-32. doi: 10.1016/j.gie.2013.04.185. Epub 2013 Jul 30. PMID 23910062
- [Background] Sano Y, Tanaka S, Kudo SE, Saito S, Matsuda T, Wada Y, Fujii T, Ikematsu H, Uraoka T, Kobayashi N, Nakamura H, Hotta K, Horimatsu T, Sakamoto N, Fu KI, Tsuruta O, Kawano H, Kashida H, Takeuchi Y, Machida H, Kusaka T, Yoshida N, Hirata I, Terai T, Yamano HO, Kaneko K, Nakajima T, Sakamoto T, Yamaguchi Y, Tamai N, Nakano N, Hayashi N, Oka S, Iwatate M, Ishikawa H, Murakami Y, Yoshida S, Saito Y. Narrow-band imaging (NBI) magnifying endoscopic classification of colorectal tumors proposed by the Japan NBI Expert Team. Dig Endosc. 2016 Jul;28(5):526-33. doi: 10.1111/den.12644. Epub 2016 Apr 20. PMID 26927367
- [Background] Puig I, Lopez-Ceron M, Arnau A, Rosinol O, Cuatrecasas M, Herreros-de-Tejada A, Ferrandez A, Serra-Burriel M, Nogales O, Vida F, de Castro L, Lopez-Vicente J, Vega P, Alvarez-Gonzalez MA, Gonzalez-Santiago J, Hernandez-Conde M, Diez-Redondo P, Rivero-Sanchez L, Gimeno-Garcia AZ, Burgos A, Garcia-Alonso FJ, Bustamante-Balen M, Martinez-Bauer E, Penas B, Pellise M; EndoCAR group, Spanish Gastroenterological Association and the Spanish Digestive Endoscopy Society. Accuracy of the Narrow-Band Imaging International Colorectal Endoscopic Classification System in Identification of Deep Invasion in Colorectal Polyps. Gastroenterology. 2019 Jan;156(1):75-87. doi: 10.1053/j.gastro.2018.10.004. Epub 2018 Oct 6. PMID 30296432